CLINICAL TRIAL: NCT01039792
Title: Double Blind Placebo Controlled Trial of Methyl B12 on Behavioral and Metabolic Measures in Children With Autism
Brief Title: Trial of Methyl B12 on Behavioral and Metabolic Measures in Children With Autism
Acronym: B12
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Davis (Other); Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Robert Hendren, Professor of Psychiatry, Director of Child & Adolescent Psychiatry, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Autism Speaks 3031
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Autistic Disorder
Keywords: Autism; Pervasive Developmental Disorders
MeSH Terms: conditions — Autistic Disorder; Child Development Disorders, Pervasive | interventions — Vitamin B 12; mecobalamin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- Active (Experimental): Active Methyl B12
  Interventions: Drug: Methyl B12

INTERVENTIONS:
Drug: Methyl B12 — 75 µg/Kg subcutaneously injected once every 3 days
  Other Names: Vitamin B12; methylcobalamin
  Arms: Active
Dietary Supplement: Placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the supplement Methyl B12 is effective in treating some of the symptoms of Autism.

DETAILED DESCRIPTION:
Autism is a complex neurodevelopmental disorder with early childhood onset characterized by impairments in communication, social interaction, and repetitive behavior. Due to the lack of known treatments for autism, many parents seek complementary and alternative medical (CAM) therapies hoping to help their affected child. Methylcobalamin (methyl B12) is a commonly used CAM treatment that has anecdotal reports of remarkable clinical improvements with few side effects. Prior studies have found that children with autism have deficiencies in key metabolites and antioxidants which can be caused by methyl B12 deficiency; additional studies have shown that methyl B12 normalizes deficiencies in these metabolites and antioxidants. Based on these reports, a pilot study was conducted at UC Davis on the effect of methyl B12 on the behavioral and metabolic measures in children with autism. The preliminary results of 29 subjects revealed a subgroup of 9 responders to clinical behavior assessments. These responders also demonstrated significant improvement on the plasma measures of antioxidant capacity, suggesting methyl B12 improves symptoms in a subgroup of children with autism by increasing key antioxidants. The current study will have an 8 week double blind design with 50 subjects, designed to evaluate improvements from methyl B12 by using behavioral assessments and analysis of specific metabolites in the subjects' blood. This study will determine whether methyl B12 will lead to benefits in any of the core features of autism, and will examine metabolic changes with the hope of potentially identifying a biomarker for treatment response in a subgroup of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DSM IV defined autism and meets cut off on Autism Diagnostic Inventory-Revised (ADI-R) and/or the Autism Diagnostic Observation Scale (ADOS)
* Age 3 through 7 years
* IQ of 50 or above
* Parental agreement to continue present dietary, behavioral or psychotropic drug treatment but not change treatment during 8 week intervention
* Willingness to have blood drawn, without the use of a sedative prescription from the study doctor

Exclusion Criteria:

* Bleeding disorder
* Cancer
* Seizure disorder
* Fragile X or other known genetic cause of autism
* Perinatal brain injury (i.e.: cerebral palsy)
* Other serious medical illnesses
* Current use of any B12 supplement

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2010-01; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Hendren, DO, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

REFERENCES:
- [Derived] Hendren RL, James SJ, Widjaja F, Lawton B, Rosenblatt A, Bent S. Randomized, Placebo-Controlled Trial of Methyl B12 for Children with Autism. J Child Adolesc Psychopharmacol. 2016 Nov;26(9):774-783. doi: 10.1089/cap.2015.0159. Epub 2016 Feb 18. PMID 26889605

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited from the Autism clinic, an advertisement on Craigslist.org and letters to families of current and previous patients, between 12/8/10 to 10/22/13.
Pre-assignment Details: Enrolled patients excluded from the trial prior to assignment phase were attributed to inattention/inability to focus, increased hyperactivity/stimming, lack of efficacy, challenging behavior- parent request to drop out
Period: Overall Study
Arm/Group | Placebo | Active
Started | 29 | 28
Completed | 23 | 27
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Population: Greater number of subjects (N=50) and thus larger power (93%), than the pilot study (N=30) was necessary to determine efficacy of methyl B12.
Groups:
- Placebo: Placebo
  Placebo: Syringes were tightly taped with opaque material to hide the color of the liquid
- Total: Total of all reporting groups
Arm/Group | Placebo | Active | Total
Number analyzed (Participants) | 23 | 27 | 50
Age, Categorical [Count of Participants; unit: Participants] — Male and female subjects between 3 and 7 years of age with a diagnosis of autism.
  Participants
    <=18 years | 23 | 27 | 50
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 58 (14) | 67 (16) | 63 (16)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 19 | 21 | 40
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 27 | 50

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression-Improvement (CGI-I)
Description: PI assesses subject's change using the CGI-I measure. This is a 7-point Likert scale that assesses improvement of the patient's condition. Scores range from the worst score of 7 (Very much worse) to the best score of 1 (Very much improved). Lower scores are better on this scale, and indicate greater improvement.
Time Frame: 8 weeks
Population: comparing placebo vs active B12 subjects
Measure: Mean (Standard Deviation); unit: CGI- Improvement
Arm/Group | Placebo | Active
Number analyzed (Participants) | 23 | 27
CGI- Improvement | 3.1 (0.8) | 2.4 (0.8)

ADVERSE EVENTS:
Arm/Group | Placebo | Active
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 14/23 | 13/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=23) | Active (N=27)
cold (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
fever (General disorders) | 1 (1) | 2 (2)
increased hyperactivity (Psychiatric disorders) | 7 (7) | 2 (2)
mouthing (General disorders) | 1 (1) | 5 (5)
trouble sleeping (General disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No